CLINICAL TRIAL: NCT05823922
Title: Feasibility and Efficacy of Mobile Cognitive Behavioral Therapy for Medical and Graduate Students
Brief Title: Mobile Cognitive Behavioral Therapy for Medical and Graduate Students
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-08025115
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Anxiety Disorders; Depression
Keywords: Anxiety; Mobile Application; Cognitive Behavioral Therapy; Graduate Students
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial designed to compare the efficacy of clinician-delivered cognitive behavior therapy supplemented with a mobile cognitive behavioral therapy program in improving anxiety and depression in graduate students. Participants will be randomized to one of two conditions: 1) Clinician-delivered Cognitive Behavior Therapy 2) Clinician-delivered Cognitive Behavior Therapy and CBT mobile app
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinician-delivered Cognitive Behavioral Therapy only (Active Comparator): Participants receive treatment with a licensed clinician for 6 weeks.
  Interventions: Behavioral: Clinician Delivered CBT
- Clinician-delivered CBT + Supplemental app (Experimental): Mobile application at least two times per week for six weeks, for at least 20 minutes on each of the two days in addition to the clinician-delivered CBT
  Interventions: Behavioral: Clinician Delivered CBT; Behavioral: Supplemental MAYA App

INTERVENTIONS:
Behavioral: Clinician Delivered CBT — Clinicians teach cognitive behavioral therapy (CBT) techniques including emotion monitoring, cognitive restructuring, mindfulness, and exposure to help individuals with anxiety and depression. Participants will attend weekly sessions with their clinician for 6 weeks.
Behavioral: Supplemental MAYA App — The Maya app teaches cognitive behavioral therapy (CBT) techniques including emotion monitoring, cognitive restructuring, mindfulness, and exposure to help individuals with anxiety.
  Participants will attend weekly sessions with their clinician as well as using the MAYA application for at least 20 minutes twice a week
  Arms: Clinician-delivered CBT + Supplemental app

SUMMARY:
The study aims to assess and compare clinician-delivered cognitive behavior therapy (CBT) supplemented with "MAYA", a mobile cognitive behavioral therapy app program to clinician-delivered cognitive behavioral therapy alone. The experimental group will be asked to use the mobile application at least two times per week for six weeks, for at least 20 minutes on each of the two days in addition to the clinician-delivered CBT. Participants will complete a weekly self-report assessment battery designed to assess anxiety and mood symptoms. The investigators think that clinician-delivered CBT supplemented with "MAYA" will improve more effective at improving symptoms of anxiety and depression than clinician-delivered CBT alone.

DETAILED DESCRIPTION:
Growing evidence suggests a need for anxiety and depression treatments that can be disseminated easily to young adults. Many do not seek out treatment for reasons including lack of availability and high cost. There is a growing need for accessible, affordable, research-supported treatments designed to increase the practice of skills and therefore improve treatment outcomes. Graduate students use mobile devices frequently; thus, mobile app-based interventions may be particularly appealing to individuals in this age range with anxiety or depression who are unable to access more traditional psychotherapy administered in person by a therapist.

The study aims to compare the efficacy and feasibility of clinician-delivered cognitive behavior therapy supplemented with the mobile app program to clinician- delivered cognitive behavioral therapy alone. Young adults with anxiety and/or depression will be randomized to clinician-delivered CBT (active control group) or to the clinician CBT + mobile app (intervention group). In the active control group, participants will participate in weekly clinician-delivered Cognitive Behavior Therapy. In the intervention group, participants will participate in weekly clinician-delivered Cognitive Behavior Therapy and use a mobile application for at least 20 minutes two times per week for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years.
* Clinically significant anxiety (as determined by a score of 10 or greater on the GAD-7) or clinically significant depression (as determined by a score of 10 or greater on the PHQ-9).
* Current graduate student at Weill Cornell Medicine.
* Access to an Apple iPhone

Exclusion Criteria:

* Lifetime diagnosis of a bipolar or psychotic disorder.
* Intent or plan to attempt suicide.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Change in anxiety symptoms from baseline to end of treatment as measured by the GAD-7. | Baseline to endpoint [Week 6]
  The primary symptom measure for anxiety will be the Generalized Anxiety Disorder 7-item scale. The GAD-7 is a 7-item self-report questionnaire measure of the severity of generalized anxiety symptoms. Scores range from 0 to 27 where higher scores indicate a greater severity of symptoms, and lower scores indicate mild to no anxiety symptoms.
Change in depressive symptoms from baseline to end of treatment as measured by the PHQ-9 | Baseline to endpoint [Week 6]
  The primary symptom measure for depression will be the Patient Health Questionnaire 9-item measure (PHQ-9). The PHQ-9 is a 9-item self-report questionnaire measure of the severity of depression symptoms. Scores range from 0 to 27, where higher scores indicate a greater severity of symptoms, and lower scores indicate mild to no depression symptoms.

SECONDARY OUTCOMES:
Adherence as measured by the mean difference in total number of completed clinician assigned homework between groups | Endpoint [Week 6]
Retention as measured by the mean difference in total number of completed study weeks between groups | Endpoint [Week 6]

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Marino, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No